CLINICAL TRIAL: NCT01631214
Title: A Multicenter, International, Randomized, Double-blind, Alendronate-controlled Study to Determine the Efficacy and Safety of Romosozumab in the Treatment of Postmenopausal Women With Osteoporosis
Brief Title: Study to Determine the Efficacy and Safety of Romosozumab in the Treatment of Postmenopausal Women With Osteoporosis
Acronym: ARCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110142; 2011-003142-41 (EudraCT Number)
Record Dates: First submitted 2012-05-24; First posted 2012-06-29 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Postmenopausal Women With Osteoporosis
Keywords: Osteoporosis, Osteoporosis-postmenopausal, Bone Diseases-Metabolic, Bone Diseases, Musculoskeletal Diseases
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal; Bone Diseases, Metabolic; Bone Diseases; Musculoskeletal Diseases | interventions — romosozumab; Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alendronate/Alendronate (Active Comparator): Participants received 70 mg alendronate once a week and placebo to romosozumab subcutaneously once a month for the first 12 months. After completion of the 12-month double-blind treatment period participants continued to receive 70 mg alendronate once a week until the end of the study.
  Interventions: Drug: Alendronate; Drug: Placebo to Romosozumab
- Romosozumab/Alendronate (Experimental): Participants received 210 mg romosozumab subcutaneously once a month and placebo to alendronate orally once a week for the first 12 months. After completion of the 12-month double-blind treatment period participants received 70 mg alendronate once a week until the end of the study.
  Interventions: Biological: Romosozumab; Drug: Alendronate; Drug: Placebo to Alendronate

INTERVENTIONS:
Biological: Romosozumab — Romosozumab 210 mg administered by subcutaneous injection once a month during the double-blind treatment phase.
  Other Names: AMG 785; Evenity
  Arms: Romosozumab/Alendronate
Drug: Alendronate — Alendronate 70 mg tablet taken once a week
  Other Names: Fosamax
Drug: Placebo to Romosozumab — Administered by subcutaneous injection once a month during the double-blind treatment phase.
  Arms: Alendronate/Alendronate
Drug: Placebo to Alendronate — Matching placebo tablet taken once a week during the double-blind treatment phase.
  Arms: Romosozumab/Alendronate

SUMMARY:
The purpose of this study is to determine if treatment is effective in preventing fractures in women with postmenopausal osteoporosis.

DETAILED DESCRIPTION:
In this trial, women were randomly assigned in a 1:1 ratio to receive monthly subcutaneous romosozumab or weekly oral alendronate for 12 months. Randomization was stratified according to age (<75 vs. ≥75 years). After completion of the double-blind treatment period, all the participants were to receive open-label weekly oral alendronate until the end of the trial, with blinding to the initial treatment assignment maintained.

The primary analysis was performed when clinical fracture events had been confirmed in at least 330 participants and all the participants had completed the month 24 visit. The study was to continue in an event-driven manner until at least 440 participants experienced a nonvertebral fracture or if the superiority of romosozumab was proven for nonvertebral fractures at the primary analysis.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women who meet at least one of the following bone mineral density (BMD) and fracture criteria:

* BMD T-score at the total hip or femoral neck of ≤ -2.50 and EITHER:

  * at least 1 moderate (semiquantitative grade [SQ]2) or severe (SQ3) vertebral fracture OR
  * at least 2 mild (SQ1) vertebral fractures OR
* BMD T-score at the total hip or femoral neck of ≤ -2.00 and EITHER:

  * at least 2 moderate (SQ2) or severe (SQ3) vertebral fractures OR
  * a fracture of the proximal femur that occurred within 3 to 24 months prior to randomization.

Exclusion Criteria:

* History of metabolic or bone disease (except osteoporosis)
* Use of agents affecting bone metabolism
* Vitamin D insufficiency
* History of solid organ or bone marrow transplants
* Hyper- or hypocalcemia
* Hyper- or hypothyroidism
* Hyper- or hypoparathyroidism
* Possible signs of intolerance to alendronate

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4093 (Actual)
Dates: Start 2012-05-04 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (255):
- United States (32):
  - Research Site, Birmingham, Alabama
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Downey, California
  - Research Site, Greenbrae, California
  - Research Site, Los Angeles, California
  - Research Site, South Lake Tahoe, California
  - Research Site, Tustin, California
  - Research Site, Walnut Creek, California
  - Research Site, Lakewood, Colorado
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Miami, Florida
  - Research Site, Stuart, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Gainesville, Georgia
  - Research Site, Maywood, Illinois
  - Research Site, Quincy, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Bethesda, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Las Cruces, New Mexico
  - Research Site, Great Neck, New York
  - Research Site, Bismarck, North Dakota
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Richmond, Virginia
  - Research Site, Port Angeles, Washington
  - Research Site, Madison, Wisconsin
- Argentina (5):
  - Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Buenos Aires
- Australia (7):
  - Research Site, Darlinghurst, New South Wales
  - Research Site, Kogarah, New South Wales
  - Research Site, Randwick, New South Wales
  - Research Site, Box Hill, Victoria
  - Research Site, Geelong, Victoria
  - Research Site, Heidelberg West, Victoria
  - Research Site, Parkville, Victoria
- Austria (3):
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (6):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (8):
  - Research Site, Fortaleza, Ceará
  - Research Site, Vitória, Espírito Santo
  - Research Site, Brasília, Federal District
  - Research Site, Goiânia, Goiás
  - Research Site, Curitiba, Paraná
  - Research Site, Recife, Pernambuco
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (10):
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Kitchener, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Westmout, Quebec
- Research Site, Santiago, Chile
- Colombia (5):
  - Research Site, Medellín, Antioquia
  - Research Site, Barranquilla, Atlántico
  - Research Site, Bogota, Cundinamarca
  - Research Site, Bogotá
  - Research Site, Bucaramanga
- Czechia (10):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Klatovy
  - Research Site, Opava
  - Research Site, Ostrava-Trebovice
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Uherské Hradiště
  - Research Site, Zlín
- Denmark (8):
  - Research Site, Aalborg
  - Research Site, Århus C
  - Research Site, Ballerup Municipality
  - Research Site, Glostrup Municipality
  - Research Site, Hvidovre
  - Research Site, Køge
  - Research Site, Odense
  - Research Site, Vejle
- Dominican Republic (3):
  - Research Site, Santo Domingo, Nacional
  - Research Site, Santiago de los Caballeros, Santiago Province
  - Research Site, Santo Domingo
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Finland (4):
  - Research Site, Helsinki
  - Research Site, Jyväskylä
  - Research Site, Kuopio
  - Research Site, Turku
- France (8):
  - Research Site, Bordeaux
  - Research Site, Cahors
  - Research Site, Lille
  - Research Site, Lyon Cédex 3
  - Research Site, Orléans
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Germany (14):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Dresden
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heinsberg
  - Research Site, Hellersdorf
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Würzburg
- Greece (3):
  - Research Site, Athens
  - Research Site, Larissa
  - Research Site, Thessaloniki
- Guatemala (2):
  - Research Site, Antigua Guatemala, Departamento de Sacatepéquez
  - Research Site, Guatemala City
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, New Territories
- Hungary (10):
  - Research Site, Balatonfüred
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Kiskunhalas
  - Research Site, Kistarcsa
  - Research Site, Veszprém
  - Research Site, Zalaegerszeg
- Ireland (3):
  - Research Site, Cork
  - Research Site, Dublin
  - Research Site, Galway
- Israel (4):
  - Research Site, Bnei Brak
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Tel Aviv
- Italy (10):
  - Research Site, Arenzano GE
  - Research Site, Bologna
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Siena
  - Research Site, Torino
  - Research Site, Verona
- Latvia (2):
  - Research Site, Liepāja
  - Research Site, Riga
- Research Site, Vilnius, Lithuania
- Mexico (7):
  - Research Site, Mexicali, Baja California Norte
  - Research Site, Mexicalli, Baja California Norte
  - Research Site, León, Guanajuato
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo León
  - Research Site, Querétaro City, Querétaro
  - Research Site, Ciudad Obregón, Sonora
- Netherlands (3):
  - Research Site, Leiden
  - Research Site, Rotterdam
  - Research Site, Venlo
- New Zealand (2):
  - Research Site, Christchurch
  - Research Site, Grafton, Auckland
- Norway (4):
  - Research Site, Elverum
  - Research Site, Hamar
  - Research Site, Oslo
  - Research Site, Stavanger
- Research Site, Lima, Peru
- Poland (14):
  - Research Site, Bialystok
  - Research Site, Dabrowka Dopiewo
  - Research Site, Elblag
  - Research Site, Gdynia
  - Research Site, Gliwice
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Świdnik
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Oradea
  - Research Site, Târgu Mureş
- Russia (8):
  - Research Site, Arkhangelsk
  - Research Site, Ivanovo
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Petrozavodsk
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Slovakia (6):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Kosice-Saca
  - Research Site, Lučenec
  - Research Site, Piešťany
  - Research Site, Trenčín
- South Africa (5):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Pretoria, Gauteng
  - Research Site, Parow, Western Cape
  - Research Site, Somerset West, Western Cape
  - Research Site, Tygerberg
- South Korea (6):
  - Research Site, Daegu
  - Research Site, Guri-si
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Suwon-si, Gyeonggi-do
- Spain (7):
  - Research Site, Granada, Andalusia
  - Research Site, Seville, Andalusia
  - Research Site, Santander, Cantabria
  - Research Site, Barcelona, Catalonia
  - Research Site, Sant Joan Despí, Catalonia
  - Research Site, A Coruña, Galicia
  - Research Site, Madrid
- Sweden (4):
  - Research Site, Linköping
  - Research Site, Mölndal
  - Research Site, Stockholm
  - Research Site, Umeå
- Taiwan (2):
  - Research Site, Tainan
  - Research Site, Taipei
- Turkey (Türkiye) (3):
  - Research Site, Adana
  - Research Site, Istanbul
  - Research Site, Izmir
- United Kingdom (15):
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, Cardiff
  - Research Site, Chorley
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Liverpool
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Norwich
  - Research Site, Reading
  - Research Site, Sheffield
  - Research Site, Sidcup
  - Research Site, Staffordshire
  - Research Site, Warwick

REFERENCES:
- [Background] Saag KG, Petersen J, Brandi ML, Karaplis AC, Lorentzon M, Thomas T, Maddox J, Fan M, Meisner PD, Grauer A. Romosozumab or Alendronate for Fracture Prevention in Women with Osteoporosis. N Engl J Med. 2017 Oct 12;377(15):1417-1427. doi: 10.1056/NEJMoa1708322. Epub 2017 Sep 11. PMID 28892457
- [Background] Cosman F, Lewiecki EM, Ebeling PR, Hesse E, Napoli N, Matsumoto T, Crittenden DB, Rojeski M, Yang W, Libanati C, Ferrari S. T-Score as an Indicator of Fracture Risk During Treatment With Romosozumab or Alendronate in the ARCH Trial. J Bone Miner Res. 2020 Jul;35(7):1333-1342. doi: 10.1002/jbmr.3996. Epub 2020 May 22. PMID 32445228
- [Background] Lau EMC, Dinavahi R, Woo YC, Wu CH, Guan J, Maddox J, Tolman C, Yang W, Shin CS. Romosozumab or alendronate for fracture prevention in East Asian patients: a subanalysis of the phase III, randomized ARCH study. Osteoporos Int. 2020 Apr;31(4):677-685. doi: 10.1007/s00198-020-05324-0. Epub 2020 Feb 11. PMID 32047951
- [Background] Miller PD, Adachi JD, Albergaria BH, Cheung AM, Chines AA, Gielen E, Langdahl BL, Miyauchi A, Oates M, Reid IR, Santiago NR, Vanderkelen M, Wang Z, Yu Z. Efficacy and Safety of Romosozumab Among Postmenopausal Women With Osteoporosis and Mild-to-Moderate Chronic Kidney Disease. J Bone Miner Res. 2022 Aug;37(8):1437-1445. doi: 10.1002/jbmr.4563. Epub 2022 May 20. PMID 35466448
- [Background] Brown JP, Engelke K, Keaveny TM, Chines A, Chapurlat R, Foldes AJ, Nogues X, Civitelli R, De Villiers T, Massari F, Zerbini CAF, Wang Z, Oates MK, Recknor C, Libanati C. Romosozumab improves lumbar spine bone mass and bone strength parameters relative to alendronate in postmenopausal women: results from the Active-Controlled Fracture Study in Postmenopausal Women With Osteoporosis at High Risk (ARCH) trial. J Bone Miner Res. 2021 Nov;36(11):2139-2152. doi: 10.1002/jbmr.4409. Epub 2021 Aug 10. PMID 34190361
- [Background] McClung MR, Betah D, Leder BZ, Kendler DL, Oates M, Timoshanko J, Wang Z. Romosozumab improves microarchitecture as assessed by tissue thickness-adjusted trabecular bone score in postmenopausal women with osteoporosis. J Bone Miner Res. 2025 Feb 2;40(2):193-200. doi: 10.1093/jbmr/zjae194. PMID 39656908
- [Background] Ferrari S, Betah D, Feldman RG, Langdahl BL, Oates M, Timoshanko J, Wang Z, Dhaliwal R. Romosozumab Improves Tissue Thickness-Adjusted Trabecular Bone Score in Women With Osteoporosis and Diabetes. J Clin Endocrinol Metab. 2025 Sep 16;110(10):2861-2868. doi: 10.1210/clinem/dgae862. PMID 39854280
- [Derived] Lane J, Langdahl B, Stone M, Kurth A, Oates M, Timoshanko J, Wang Z, Libanati C, Cosman F. Romosozumab in patients who experienced an on-study fracture: post hoc analyses of the FRAME and ARCH phase 3 trials. Osteoporos Int. 2024 Jul;35(7):1195-1204. doi: 10.1007/s00198-024-07049-w. Epub 2024 Apr 4. PMID 38573517
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 270 centers in 41 countries globally from 04 May 2012 to 29 June 2017.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive romosozumab or alendronate for 12 months. Randomization was stratified by age (< 75 vs. ≥ 75 years). After completion of the double-blind trial period, all participants received open-label alendronate until the end of the trial, with blinding to the initial treatment assignment maintained.
Period: Overall Study
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Started | 2047 | 2046
Received Double-blind Treatment | 2040 | 2038
Completed Double-blind Period (Completion of the double-blind period is defined as having attended the month 12 study visit.) | 1823 | 1831
Completed Primary Analysis Period (Completion of the primary analysis period is defined as ongoing at the primary analysis cutoff date.) | 1576 | 1574
Completed | 1503 | 1523
Not Completed | 544 | 523
Not completed — Withdrawal by Subject | 276 | 290
Not completed — Death | 113 | 106
Not completed — Lost to Follow-up | 54 | 40
Not completed — Adverse Event | 45 | 45
Not completed — Other | 22 | 19
Not completed — Noncompliance | 16 | 15
Not completed — Requirement for Alternative Therapy | 8 | 3
Not completed — Protocol Deviation | 4 | 3
Not completed — Ineligibility determined | 5 | 2
Not completed — Administrative Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate | Total
Number analyzed (Participants) | 2047 | 2046 | 4093
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (7.5) | 74.4 (7.5) | 74.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2047 | 2046 | 4093
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 662 | 631 | 1293
  Not Hispanic or Latino | 1385 | 1415 | 2800
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 5 | 12
  Asian | 149 | 137 | 286
  Black or African American | 23 | 19 | 42
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  White | 1415 | 1447 | 2862
  Multiple | 4 | 2 | 6
  Other | 446 | 436 | 882
  Missing | 1 | 0 | 1
Age Strata per Randomization [Count of Participants; unit: Participants]
  < 75 years | 976 | 973 | 1949
  ≥ 75 years | 1071 | 1073 | 2144
Severe Vertebral Fracture [Count of Participants; unit: Participants] — A participant had a prevalent vertebral fracture if any vertebra from T4 to L4 had a grade of 3 at baseline based on an assessment of spinal radiographs using the Genant Semiquantitative Scoring Method. A grade 3 fracture is defined as approximately 40% or greater reduction in anterior, middle, and/or posterior height.
  Participants
    Presence | 1321 | 1369 | 2690
    Absence | 726 | 677 | 1403
Total Hip Bone Mineral Density (BMD) T-score [Count of Participants; unit: Participants] — BMD was measured using dual-energy x-ray absorptiometry (DXA). The T-score is a comparison of a person's bone density with that of a healthy 30-year-old of the same sex. Lower scores (more negative) mean lower bone density: A T-score of -2.5 or lower qualifies as osteoporosis and a T-score of -1.0 to - 2.5 signifies osteopenia, meaning below-normal bone density without full osteoporosis.
  Participants
    ≤ -2.5 | 1384 | 1356 | 2740
    > -2.5 | 662 | 690 | 1352
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With New Vertebral Fractures Through Month 24
Description: All fracture assessments were performed by blinded central imaging readers.
  New vertebral fractures occurred when there was ≥ 1 grade increase from the previous grade of 0 in any vertebra from T4 to L4 using the Genant Semiquantitative Scoring method based on assessment of x-rays according to the following scale:
  * Grade 0 (Normal) = no fracture;
  * Grade 1 (Mild) = mild fracture, 20 to 25% reduction in vertebral height (anterior, middle, or posterior);
  * Grade 2 (Moderate) = moderate fracture, 25 to 40% reduction in anterior, middle, and/or posterior height;
  * Grade 3 (Severe) = severe fracture, greater than 40% reduction in anterior, middle, and/or posterior height.
  Incident vertebral fractures were confirmed by a second independent reader using the Semiquantitative method.
Time Frame: 24 months
Population: Randomized participants with a baseline and ≥ 1 postbaseline evaluation of vertebral fracture, including participants who had vertebrae with missing Genant semiquantitative scores at baseline whose first postbaseline spinal radiograph showed no fracture on the same vertebrae. Last observation carried forward imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 1834 | 1825
percentage of participants | 8.0 | 4.1
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — The primary endpoints were tested at the 5% level (2-sided), accounting for multiplicity using the Hochberg procedure. If the larger of the 2 p-values was significant at the 0.05 level (2-sided), the statistical testing continued to the secondary endpoint in the testing sequence; p < 0.001, Regression, Logistic; Based on a logistic regression model adjusted for age strata, baseline total hip BMD T-score and presence of severe vertebral fracture at baseline; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.36 to 0.64], Standard Error of Mean 0.15 — Values < 1 for odds ratio favor romosozumab. The standard error (SE) represents the standard error of log(odds ratio)
Statistical Analysis 2: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; The risk ratio (ratio of percentages, Romosozumab:Alendronate) was based on the Mantel Haenszel method, adjusted for age strata (<75 vs. ≥75 years), the presence or absence of severe vertebral fracture at baseline, and baseline bone mineral density T-score at the total hip (≤ -2.5, > -2.5). Values < 1 for risk ratio favor romosozumab; Test type: Superiority; Risk Ratio (RR) = 0.50, 95% CI 2-sided [0.38 to 0.66], Standard Error of Mean 0.14 — SE represents the standard error of log (risk ratio)
Statistical Analysis 3: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; The absolute risk reduction (difference in percentages, Alendronate - Romosozumab) was based on the Mantel-Haenszel method adjusted for age strata, baseline total hip BMD T-score (≤ -2.5, > -2.5), and presence of severe vertebral fracture at baseline. Positive values for absolute risk reduction favor romosozumab; Test type: Superiority; Absolute risk reduction = 4.03, 95% CI 2-sided [2.50 to 5.57], Standard Error of Mean 0.78

2. Primary Outcome: Percentage of Participants With a Clinical Fracture at the Primary Analysis
Description: All fracture assessments were performed by blinded central imaging readers. Clinical fractures included clinical vertebral and nonvertebral fractures (excluding skull, facial, mandible, cervical vertebrae, thoracic vertebrae, lumbar vertebrae, metacarpus, finger phalanges, and toe phalanges) that were associated with signs and/or symptoms indicative of a fracture. Clinical vertebral fractures were included regardless of trauma severity or pathologic fractures; nonvertebral fractures associated with high trauma severity or pathologic fractures were excluded.
Time Frame: The primary analysis was performed when clinical fracture events had been confirmed in at least 330 patients and all participants had completed the month 24 visit. The median follow-up was 2.7 years (interquartile range, 2.2 to 3.3).
Population: All randomized participants. Missing values for clinical fractures were imputed using last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 13.0 | 9.7
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.61 to 0.88], Standard Error of Mean 0.09 — Hazard ratio < 1 favors romosozumab; SE represents the standard error of log (hazard ratio)

3. Secondary Outcome: Percentage of Participants With a Nonvertebral Fracture at the Primary Analysis
Description: A nonvertebral fracture was defined as a documented fracture excluding skull, facial, mandible, cervical vertebrae, thoracic vertebrae, lumbar vertebrae, metacarpus, finger phalanges, and toe phalanges. In addition, fractures associated with high trauma severity or pathologic fractures were excluded.
Time Frame: as for outcome 2
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 10.6 | 8.7
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — If the 2 primary endpoints and the specified BMD secondary endpoints were all significant, the nonvertebral fracture at the primary analysis was evaluated based on a 1-sided test (overall α=0.025) determined by the Lan-DeMets alpha spending function that approximates a Pocock boundary, 0.0233 (1-sided); p = 0.040, Regression, Cox — The adjusted 2-sided p-value is reported; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.66 to 0.99], Standard Error of Mean 0.10 — Based on Cox proportional hazards model adjusting for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline. Hazard ratio < 1 favors romosozumab; SE represents the standard error of log (hazard ratio)

4. Secondary Outcome: Percentage of Participants With Any Fracture at the Primary Analysis
Description: All fractures include any osteoporotic nonvertebral fractures that are not associated with high trauma severity or pathologic fractures and new or worsening vertebral fractures regardless of trauma severity or pathologic fractures.
Time Frame: as for outcome 2
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 19.1 | 13.0
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — This endpoint was not included in the sequential testing procedure and was analyzed without multiplicity adjustment at a significance level of 0.05 (two-sided); p < 0.001, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.56 to 0.76], Standard Error of Mean 0.08 — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Percentage of Participants With a New or Worsening Vertebral Fracture Through Month 24
Description: A new or worsening vertebral fracture was identified when there was a ≥ 1 grade increase from the previous grade in any vertebra from T4 to L4 according to the Genant Semiquantitative Scoring method based on assessment of x-rays according to the following scale:
  * Grade 0 (Normal) = no fracture;
  * Grade 1 (Mild) = mild fracture, 20 to 25% reduction in vertebral height (anterior, middle, or posterior);
  * Grade 2 (Moderate) = moderate fracture, 25 to 40% reduction in anterior, middle, and/or posterior height;
  * Grade 3 (Severe) = severe fracture, greater than 40% reduction in anterior, middle, and/or posterior height.
  Incident vertebral fractures were confirmed by a second independent reader using the Semiquantitative method.
Time Frame: 24 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 1834 | 1825
percentage of participants | 9.2 | 4.8
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Regression, Logistic; Based on logistic regression model adjusted for age strata, baseline total hip BMD T-score and presence of severe vertebral fracture at baseline; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.37 to 0.64], Standard Error of Mean 0.14 — Values < 1 for odds ratio favor romosozumab. The standard error (SE) represents the standard error of log(odds ratio)
Statistical Analysis 2: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.52, 95% CI 2-sided [0.40 to 0.66], Standard Error of Mean 0.13 — SE represents the standard error of log (risk ratio)
Statistical Analysis 3: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Absolute risk reduction = 4.44, 95% CI 2-sided [2.80 to 6.08], Standard Error of Mean 0.84

6. Secondary Outcome: Percentage of Participants With a Major Nonvertebral Fracture at the Primary Analysis
Description: Major nonvertebral fractures included a subset of nonvertebral fractures including pelvis, distal femur (ie, femur excluding hip), proximal tibia (ie, tibia excluding ankle), ribs, proximal humerus (ie, humerus excluding elbow), forearm, and hip.
Time Frame: as for outcome 2
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 9.6 | 7.1
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.004, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.59 to 0.90], Standard Error of Mean 0.11 — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Percentage of Participants With a Hip Fracture at the Primary Analysis
Description: Hip fractures were defined as a subset of nonvertebral fractures including fractures of the femur neck, femur intertrochanter, and femur subtrochanter.
Time Frame: as for outcome 2
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 3.2 | 2.0
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.015, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.42 to 0.92], Standard Error of Mean 0.20 — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Percentage of Participants With Multiple New or Worsening Vertebral Fractures Through Month 24
Description: A new or worsening vertebral fracture was identified when there was a ≥ 1 grade increase from the previous grade in any vertebra from T4 to L4 according to the Genant Semiquantitative Scoring method. A participant had multiple new or worsening vertebral fractures when there were ≥ 2 vertebrae from T4 to L4 with ≥ 1 grade increase from the previous grade. The multiple new or worsening vertebral fractures need not have occurred at the same visit. Incident vertebral fractures were confirmed by a second independent reader.
Time Frame: 24 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 1834 | 1825
percentage of participants | 2.5 | 1.3
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.008, Regression, Logistic; [statistical method as in outcome 5, analysis 1]; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.31 to 0.85], Standard Error of Mean 0.25 — Values < 1 for odds ratio favor romosozumab. The standard error (SE) represents the standard error of log(odds ratio)
Statistical Analysis 2: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.52, 95% CI 2-sided [0.32 to 0.85], Standard Error of Mean 0.25 — SE represents the standard error of log (risk ratio)
Statistical Analysis 3: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Absolute risk reduction = 1.21, 95% CI 2-sided [0.33 to 2.10], Standard Error of Mean 0.45

9. Secondary Outcome: Percentage of Participants With a Clinical Fracture Through Month 24
Description: Clinical fractures included clinical vertebral and nonvertebral fractures (excluding skull, facial, mandible, cervical vertebrae, thoracic vertebrae, lumbar vertebrae, metacarpus, finger phalanges, and toe phalanges) that were associated with signs and/or symptoms indicative of a fracture. Clinical vertebral fractures were included regardless of trauma severity or pathologic fractures; nonvertebral fractures associated with high trauma severity or pathologic fractures were excluded.
Time Frame: 24 months
Population: All randomized participants; Missing values for clinical fractures were imputed using last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 9.6 | 7.1
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.005, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.59 to 0.91], Standard Error of Mean 0.11 — [estimate comment as in outcome 3, analysis 1]

10. Secondary Outcome: Percentage of Participants With a Nonvertebral Fracture Through Month 24
Description: as for outcome 3
Time Frame: 24 months
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 7.8 | 6.3
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.074, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.64 to 1.02], Standard Error of Mean 0.12 — [estimate comment as in outcome 3, analysis 1]

11. Secondary Outcome: Percentage of Participants With a Hip Fracture Through Month 24
Description: as for outcome 7
Time Frame: 24 months
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 2.1 | 1.5
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.17, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.46 to 1.15], Standard Error of Mean 0.24 — [estimate comment as in outcome 3, analysis 1]

12. Secondary Outcome: Percentage of Participants With a Clinical Vertebral Fracture Through Month 24
Description: A clinical vertebral fracture is a new or worsening vertebral fracture assessed at either a scheduled or unscheduled visit and associated with any signs and/or symptoms of back pain indicative of a fracture, regardless of trauma severity or whether it is pathologic.
Time Frame: 24 months
Population: All randomized participants; Last observation carried forward imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 2.1 | 0.9
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.24 to 0.71], Standard Error of Mean 0.28 — [estimate comment as in outcome 3, analysis 1]

13. Secondary Outcome: Percentage of Participants With a Clinical Fracture Through Month 12
Description: as for outcome 9
Time Frame: 12 months
Population: All randomized participants; Missing values for clinical fractures were imputed using last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 5.4 | 3.9
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.027, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.54 to 0.96], Standard Error of Mean 0.15 — [estimate comment as in outcome 3, analysis 1]

14. Secondary Outcome: Percentage of Participants With New Vertebral Fractures Through Month 12
Description: New vertebral fractures occurred when there was ≥ 1 grade increase from the previous grade of 0 in any vertebra from T4 to L4 using the Genant Semiquantitative Scoring method based on assessment of x-rays according to the following scale:
  * Grade 0 (Normal) = no fracture;
  * Grade 1 (Mild) = mild fracture, 20 to 25% reduction in vertebral height (anterior, middle, or posterior);
  * Grade 2 (Moderate) = moderate fracture, 25 to 40% reduction in anterior, middle, and/or posterior height;
  * Grade 3 (Severe) = severe fracture, greater than 40% reduction in anterior, middle, and/or posterior height.
  Incident vertebral fractures were confirmed by a second independent reader.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 1703 | 1696
percentage of participants | 5.0 | 3.2
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.008, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.44 to 0.89], Standard Error of Mean 0.18 — Values < 1 for odds ratio favor romosozumab. The standard error (SE) represents the standard error of log(odds ratio)
Statistical Analysis 2: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.64, 95% CI 2-sided [0.46 to 0.89], Standard Error of Mean 0.17 — SE represents the standard error of log (risk ratio)
Statistical Analysis 3: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Absolute risk reduction = 1.84, 95% CI 2-sided [0.51 to 3.17], Standard Error of Mean 0.68

15. Secondary Outcome: Percentage of Participants With Any Fracture Through Month 12
Description: as for outcome 4
Time Frame: 12 months
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 9.2 | 6.5
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.002, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.57 to 0.88], Standard Error of Mean 0.11 — [estimate comment as in outcome 3, analysis 1]

16. Secondary Outcome: Percentage of Participants With a Nonvertebral Fracture Through Month 12
Description: A nonvertebral fracture was defined as a fracture present on a copy of radiographs or other diagnostic images such as computerized tomography (CT) or magnetic resonance imaging confirming the fracture within 14 days of reported fracture image date recorded by the study site, and/or documented in a copy of the radiology report, surgical report, or discharge summary, excluding skull, facial, mandible, cervical vertebrae, thoracic vertebrae, lumbar vertebrae, metacarpus, finger phalanges, and toe phalanges. In addition, fractures associated with high trauma severity or pathologic fractures were excluded.
Time Frame: 12 months
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 4.6 | 3.4
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.057, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.54 to 1.01], Standard Error of Mean 0.16 — [estimate comment as in outcome 3, analysis 1]

17. Secondary Outcome: Percentage of Participants With a Hip Fracture Through Month 12
Description: as for outcome 7
Time Frame: 12 months
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 1.1 | 0.7
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.19, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.33 to 1.26], Standard Error of Mean 0.34 — [estimate comment as in outcome 3, analysis 1]

18. Secondary Outcome: Percentage of Participants With a Major Osteoporotic Fracture Through Month 12
Description: Major osteoporotic fractures included clinical vertebral fractures and fractures of the hip, forearm and humerus. Fractures associated with high trauma severity or pathologic fractures were excluded.
Time Frame: 12 months
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 4.2 | 3.0
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.053, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.52 to 1.01], Standard Error of Mean 0.17 — [estimate comment as in outcome 3, analysis 1]

19. Secondary Outcome: Percentage of Participants With a Clinical Vertebral Fracture Through Month 12
Description: as for outcome 12
Time Frame: 12 months
Population: All randomized participants; Last observation carried forward imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 2047 | 2046
percentage of participants | 0.9 | 0.5
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.14, Regression, Cox; Model adjusted for age strata, baseline total hip BMD T-score, and presence of severe vertebral fracture at baseline; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.26 to 1.22], Standard Error of Mean 0.39 — [estimate comment as in outcome 3, analysis 1]

20. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Lumbar Spine at Month 24
Description: Bone mineral density (BMD) was measured by dual-energy x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center.
Time Frame: Baseline and month 24
Population: All randomized participants with a baseline and ≥ 1 post-baseline evaluation during the open-label period at or before month 24; Missing values were imputed by carrying forward the last non-missing post-baseline value in the open-label treatment period prior to the missing value.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 1577 | 1571
percent change | 7.2 (0.2) | 15.3 (0.2)
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Between-group comparisons of the percent change from baseline in bone mineral density were analyzed using an analysis of covariance (ANCOVA) model adjusted for treatment, age strata, presence of severe vertebral fracture at baseline, baseline BMD value, machine type, and baseline BMD value-by-machine type interaction; Test type: Superiority — If the differences in both primary end points were significant with the use of the Hochberg procedure, a fixed-sequence testing procedure was used for bone mineral density and the key secondary end point of nonvertebral fracture to adjust for multiple comparisons and to maintain an overall significance level of 0.05; p < 0.001, ANCOVA; LS Mean Difference = 8.1, 95% CI 2-sided [7.58 to 8.57], Standard Error of Mean 0.3

21. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Total Hip at Month 24
Description: as for outcome 20
Time Frame: Baseline and month 24
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 1627 | 1622
percent change | 3.5 (0.1) | 7.2 (0.1)
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; Between-group comparisons of the percent change from baseline in bone mineral density were analyzed using an ANCOVA model adjusted for treatment, age strata, presence of severe vertebral fracture at baseline, baseline BMD value, machine type, and baseline BMD value-by-machine type interaction; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p < 0.001, ANCOVA; LS Mean Difference = 3.8, 95% CI 2-sided [3.42 to 4.10], Standard Error of Mean 0.2

22. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Femoral Neck at at Month 24
Description: as for outcome 20
Time Frame: Baseline and month 24
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 1627 | 1622
percent change | 2.3 (0.2) | 6.0 (0.2)
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; [analysis description as in outcome 21, analysis 1]; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p < 0.001, ANCOVA; LS Mean Difference = 3.8, 95% CI 2-sided [3.40 to 4.14], Standard Error of Mean 0.2

23. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Lumbar Spine at Month 12
Description: as for outcome 20
Time Frame: Baseline and month 12
Population: All randomized participants with a baseline and ≥ 1 post-baseline evaluation at or before month 12; Last observation carried forward imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 1718 | 1722
percent change | 5.0 (0.1) | 13.7 (0.2)
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; [analysis description as in outcome 21, analysis 1]; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p < 0.001, ANCOVA; LS Mean Difference = 8.7, 95% CI 2-sided [8.31 to 9.09], Standard Error of Mean 0.2

24. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Total Hip at Month 12
Description: as for outcome 20
Time Frame: Baseline and month 12
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 1781 | 1781
percent change | 2.8 (0.1) | 6.2 (0.1)
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; [analysis description as in outcome 21, analysis 1]; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p < 0.001, ANCOVA; LS Mean Difference = 3.3, 95% CI 2-sided [3.03 to 3.60], Standard Error of Mean 0.1

25. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Femoral Neck at Month 12
Description: as for outcome 20
Time Frame: Baseline and month 12
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 1781 | 1781
percent change | 1.7 (0.1) | 4.9 (0.1)
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; [analysis description as in outcome 21, analysis 1]; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p < 0.001, ANCOVA; LS Mean Difference = 3.2, 95% CI 2-sided [2.90 to 3.54], Standard Error of Mean 0.2

26. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Lumbar Spine at Month 36
Description: as for outcome 20
Time Frame: Baseline and month 36
Population: All randomized participants with a baseline and ≥ 1 post-baseline evaluation during the open-label period at or before month 36; Missing values were imputed by carrying forward the last non-missing post-baseline value in the open-label treatment period prior to the missing value.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 1597 | 1593
percent change | 7.8 (0.2) | 15.2 (0.2)
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; [analysis description as in outcome 21, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, ANCOVA; LS Mean Difference = 7.4, 95% CI 2-sided [6.84 to 7.89], Standard Error of Mean 0.3

27. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Total Hip at Month 36
Description: as for outcome 20
Time Frame: Baseline and month 36
Population: as for outcome 26
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 1653 | 1653
percent change | 3.5 (0.1) | 7.2 (0.1)
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; [analysis description as in outcome 21, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, ANCOVA; LS Mean Difference = 3.7, 95% CI 2-sided [3.29 to 4.02], Standard Error of Mean 0.2

28. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Femoral Neck at Month 36
Description: as for outcome 20
Time Frame: Baseline and month 36
Population: as for outcome 26
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alendronate/Alendronate | Romosozumab/Alendronate
Number analyzed (Participants) | 1653 | 1653
percent change | 2.4 (0.2) | 6.0 (0.2)
Statistical Analysis 1: Comparison: Alendronate/Alendronate vs Romosozumab/Alendronate; [analysis description as in outcome 21, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, ANCOVA; LS Mean Difference = 3.6, 95% CI 2-sided [3.18 to 3.97], Standard Error of Mean 0.2

ADVERSE EVENTS:
Time Frame: Double-blind treatment phase: 12 months. Overall study period: From first dose of study drug up to the end of study for participants who received at any open-label dose and up to the end of the double-blind period for participants who did not. The median duration of follow-up time was 36 months.
Description: The safety analysis set included all randomized subjects who received ≥ 1 active dose of investigational product in the 12-month double-blind alendronate-controlled study period. Two participants randomized to alendronate received romosozumab in error and are counted in the romosozumab group for safety.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Double-blind Period: Alendronate 70 mg QW: Participants received 70 mg alendronate once a week (QW) and placebo to romosozumab subcutaneously once a month for 12 months during the double-blind treatment period.
- Double-blind Period: Romosozumab 210 mg QM: Participants received 210 mg romosozumab subcutaneously once a month (QM) and placebo to alendronate orally once a week for the first 12 months during the double-blind treatment period.
- Overall Study: Alendronate / Alendronate: Participants received 70 mg alendronate once a week and placebo to romosozumab subcutaneously once a month for the first 12 months. After completion of the 12-month double-blind treatment period participants continued to receive 70 mg alendronate once a week until the end of the study.
- Overall Study: Romosozumab / Alendronate: Participants received 210 romosozumab mg subcutaneously once a month and placebo to alendronate orally once a week for the first 12 months. After completion of the 12-month double-blind treatment period participants received 70 mg alendronate once a week until the end of the study.
Arm/Group | Double-blind Period: Alendronate 70 mg QW | Double-blind Period: Romosozumab 210 mg QM | Overall Study: Alendronate / Alendronate | Overall Study: Romosozumab / Alendronate
All-Cause Mortality (participants affected / at risk) | 22/2014 | 30/2040 | 103/2014 | 101/2040
Serious Adverse Events (participants affected / at risk) | 278/2014 | 262/2040 | 638/2014 | 611/2040
Other Adverse Events (participants affected / at risk) | 1190/2014 | 1112/2040 | 1498/2014 | 1424/2040
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Period: Alendronate 70 mg QW (N=2014) | Double-blind Period: Romosozumab 210 mg QM (N=2040) | Overall Study: Alendronate / Alendronate (N=2014) | Overall Study: Romosozumab / Alendronate (N=2040)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 9 | 7
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1 | 4 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 2 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 8 | 15 | 16
Angina pectoris (Cardiac disorders) | 3 | 2 | 6 | 7
Angina unstable (Cardiac disorders) | 2 | 2 | 7 | 5
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 2
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 1 | 2
Arteriospasm coronary (Cardiac disorders) | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 3 | 17 | 12
Atrial flutter (Cardiac disorders) | 0 | 1 | 1 | 2
Atrioventricular block complete (Cardiac disorders) | 3 | 0 | 4 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2 | 2
Cardiac disorder (Cardiac disorders) | 0 | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 5 | 5 | 25 | 18
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 2
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 5 | 1
Cardiac failure congestive (Cardiac disorders) | 5 | 2 | 12 | 9
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 2 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 2 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 3
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 1 | 3 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 5 | 3
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 1 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0 | 2 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial fibrosis (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 5 | 8 | 8
Myocardial ischaemia (Cardiac disorders) | 1 | 3 | 4 | 6
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 2
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 5 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 2 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 2 | 5
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vestibular ataxia (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Basedow's disease (Endocrine disorders) | 1 | 0 | 1 | 1
Goitre (Endocrine disorders) | 2 | 0 | 4 | 1
Hypercorticoidism (Endocrine disorders) | 0 | 0 | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 1
Toxic goitre (Endocrine disorders) | 0 | 0 | 0 | 1
Amaurosis (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 4 | 3 | 9 | 11
Diplopia (Eye disorders) | 0 | 1 | 0 | 1
Endocrine ophthalmopathy (Eye disorders) | 1 | 0 | 1 | 1
Entropion (Eye disorders) | 0 | 0 | 0 | 1
Glaucoma (Eye disorders) | 1 | 0 | 1 | 1
Macular fibrosis (Eye disorders) | 0 | 1 | 0 | 2
Neovascular age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 1
Retinal artery thrombosis (Eye disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 1 | 0
Vitreous prolapse (Eye disorders) | 0 | 0 | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 2 | 2 | 2
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 3
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 3 | 6
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 1 | 3 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Duodenal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Femoral hernia incarcerated (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 1 | 3 | 4
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 6 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 6
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Ileus (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 4 | 2
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 2 | 4
Intestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 2 | 2
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Mesenteric arterial occlusion (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2 | 2 | 2
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3 | 0 | 5
Volvulus (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 3
Adverse event (General disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 1 | 3
Chest pain (General disorders) | 0 | 2 | 2 | 3
Death (General disorders) | 2 | 1 | 21 | 14
Feeling abnormal (General disorders) | 1 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 2 | 2
Hypothermia (General disorders) | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 2 | 0
Malaise (General disorders) | 1 | 1 | 1 | 2
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 2 | 3
Non-cardiac chest pain (General disorders) | 2 | 1 | 4 | 1
Oedema peripheral (General disorders) | 1 | 0 | 2 | 1
Pain (General disorders) | 0 | 1 | 1 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Strangulated hernia (General disorders) | 0 | 0 | 1 | 0
Sudden death (General disorders) | 2 | 1 | 4 | 6
Ulcer haemorrhage (General disorders) | 0 | 0 | 0 | 1
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 1 | 0
Ampulla of Vater stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 1 | 1 | 1
Biliary cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Biliary fibrosis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 3 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1 | 3 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 6 | 5 | 9 | 7
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 2
Amyloidosis (Immune system disorders) | 1 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 3 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 1 | 8 | 11
Bronchitis bacterial (Infections and infestations) | 1 | 0 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 3 | 1 | 6 | 5
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 1 | 1
Dermatitis infected (Infections and infestations) | 1 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 1 | 6
Empyema (Infections and infestations) | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 2 | 2
Escherichia sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1
Gastritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 2 | 6 | 5
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 2
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 1
Haematoma infection (Infections and infestations) | 0 | 0 | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 2 | 1
Infected bite (Infections and infestations) | 0 | 0 | 0 | 1
Infected fistula (Infections and infestations) | 1 | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 2 | 3
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 1
Nosocomial infection (Infections and infestations) | 0 | 1 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 0 | 1
Pancreas infection (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 3 | 0 | 3
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 17 | 16 | 46 | 54
Pneumonia bacterial (Infections and infestations) | 3 | 1 | 6 | 4
Post procedural infection (Infections and infestations) | 1 | 0 | 1 | 1
Post procedural sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 2 | 1 | 3 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0 | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 3 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 1 | 1
Pyoderma (Infections and infestations) | 1 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 3
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 3 | 3
Septic shock (Infections and infestations) | 0 | 1 | 2 | 2
Sialoadenitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1 | 1 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 4
Urinary tract infection (Infections and infestations) | 8 | 8 | 21 | 21
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 2 | 3 | 4
Viral diarrhoea (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 1 | 2
Wound infection (Infections and infestations) | 1 | 0 | 2 | 0
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 7 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 3
Fall (Injury, poisoning and procedural complications) | 4 | 2 | 11 | 13
Femoral neck fracture (Injury, poisoning and procedural complications) | 12 | 5 | 31 | 15
Femur fracture (Injury, poisoning and procedural complications) | 12 | 11 | 51 | 42
Fibula fracture (Injury, poisoning and procedural complications) | 4 | 3 | 9 | 5
Foot fracture (Injury, poisoning and procedural complications) | 3 | 0 | 5 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Graft complication (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 7 | 3 | 16 | 6
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 8 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 2 | 5 | 6
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Pubis fracture (Injury, poisoning and procedural complications) | 4 | 0 | 7 | 3
Radius fracture (Injury, poisoning and procedural complications) | 12 | 8 | 20 | 14
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subarachnoid haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 4
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 5 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 5 | 3 | 8 | 6
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 6 | 3 | 11 | 5
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Carcinoembryonic antigen increased (Investigations) | 0 | 0 | 0 | 1
Coagulation time prolonged (Investigations) | 0 | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 1 | 0
Heart rate decreased (Investigations) | 0 | 1 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1
Medical observation normal (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 4 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3 | 7 | 7
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 2 | 17 | 11
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1 | 5 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 6 | 11 | 19
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4 | 3
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Bladder squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 4 | 5
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Cervix carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 3
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colorectal carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Epithelioid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hepatobiliary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Intra-abdominal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Lung adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 3
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 1
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Non-Hodgkin's lymphoma unspecified histology indolent stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 3
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 3
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 1 | 1
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 1
Carotid aneurysm rupture (Nervous system disorders) | 0 | 0 | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 1 | 4
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 2
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 0 | 0 | 2
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 1 | 2
Cerebral infarction (Nervous system disorders) | 0 | 0 | 2 | 3
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 3 | 1
Cerebrovascular accident (Nervous system disorders) | 7 | 6 | 15 | 19
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 2 | 2
Dementia (Nervous system disorders) | 0 | 0 | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 7 | 9
Embolic stroke (Nervous system disorders) | 0 | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 3 | 2 | 5
Essential tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0 | 2 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 2 | 0 | 4
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 2
Hypokinesia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypotonia (Nervous system disorders) | 1 | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 2 | 0 | 3 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 2 | 1 | 3
Ischaemic neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 3 | 2 | 10 | 10
Loss of consciousness (Nervous system disorders) | 0 | 0 | 2 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 2 | 1
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 1
Mixed dementia (Nervous system disorders) | 0 | 0 | 1 | 0
Monoparesis (Nervous system disorders) | 1 | 0 | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 1 | 0
Nerve root compression (Nervous system disorders) | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 1 | 1 | 1
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 2
Paresis (Nervous system disorders) | 0 | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1 | 1 | 1
Post-traumatic epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 2 | 0 | 3 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 1 | 1
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 1
Stroke in evolution (Nervous system disorders) | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 4 | 2 | 10 | 5
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 6 | 5 | 11
Vascular encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 0 | 3
Device breakage (Product Issues) | 0 | 1 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 1 | 1
Device failure (Product Issues) | 0 | 0 | 1 | 1
Device malfunction (Product Issues) | 1 | 0 | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 2
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 1 | 1 | 5 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0
Hypomania (Psychiatric disorders) | 0 | 1 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 5 | 2 | 9
Bladder prolapse (Renal and urinary disorders) | 0 | 1 | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 3 | 0 | 3 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 1
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 2
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 2 | 2
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urethral polyp (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Colpocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 2 | 2
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 2 | 2 | 2
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 2
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 3 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 6 | 5
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 | 5 | 29 | 24
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 5 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 2
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 1
Limb prosthesis user (Social circumstances) | 0 | 0 | 1 | 0
Loss of personal independence in daily activities (Social circumstances) | 0 | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1 | 0 | 2
Surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1
Umbilical hernia repair (Surgical and medical procedures) | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 1 | 4 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1 | 0 | 2
Aortic arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 2
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 2
Aortic stenosis (Vascular disorders) | 1 | 1 | 1 | 2
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1
Blood pressure inadequately controlled (Vascular disorders) | 0 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 1 | 1 | 3
Deep vein thrombosis (Vascular disorders) | 5 | 2 | 9 | 4
Embolism arterial (Vascular disorders) | 1 | 0 | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 4 | 1 | 8 | 8
Hypertensive crisis (Vascular disorders) | 2 | 0 | 5 | 1
Hypertensive emergency (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 1 | 4
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 1 | 2
Intermittent claudication (Vascular disorders) | 1 | 0 | 1 | 0
Labile hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 2 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 2 | 5 | 3
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 1 | 3 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 1
Subclavian artery occlusion (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0 | 2 | 2
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Period: Alendronate 70 mg QW (N=2014) | Double-blind Period: Romosozumab 210 mg QM (N=2040) | Overall Study: Alendronate / Alendronate (N=2014) | Overall Study: Romosozumab / Alendronate (N=2040)
Anaemia (Blood and lymphatic system disorders) | 49 | 41 | 113 | 84
Cataract (Eye disorders) | 32 | 46 | 97 | 105
Abdominal pain upper (Gastrointestinal disorders) | 63 | 62 | 109 | 101
Constipation (Gastrointestinal disorders) | 92 | 75 | 133 | 120
Diarrhoea (Gastrointestinal disorders) | 93 | 99 | 168 | 165
Gastritis (Gastrointestinal disorders) | 59 | 53 | 101 | 92
Bronchitis (Infections and infestations) | 100 | 88 | 187 | 176
Influenza (Infections and infestations) | 57 | 49 | 119 | 105
Upper respiratory tract infection (Infections and infestations) | 132 | 130 | 226 | 205
Urinary tract infection (Infections and infestations) | 128 | 97 | 244 | 180
Viral upper respiratory tract infection (Infections and infestations) | 233 | 217 | 406 | 388
Contusion (Injury, poisoning and procedural complications) | 71 | 51 | 161 | 115
Fall (Injury, poisoning and procedural complications) | 151 | 127 | 342 | 287
Arthralgia (Musculoskeletal and connective tissue disorders) | 193 | 165 | 380 | 343
Back pain (Musculoskeletal and connective tissue disorders) | 221 | 184 | 395 | 330
Muscle spasms (Musculoskeletal and connective tissue disorders) | 81 | 70 | 128 | 121
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 83 | 70 | 155 | 145
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 111 | 113 | 206 | 189
Pain in extremity (Musculoskeletal and connective tissue disorders) | 129 | 121 | 253 | 230
Dizziness (Nervous system disorders) | 80 | 85 | 152 | 149
Headache (Nervous system disorders) | 110 | 106 | 190 | 163
Cough (Respiratory, thoracic and mediastinal disorders) | 55 | 74 | 118 | 147
Hypertension (Vascular disorders) | 130 | 113 | 232 | 233

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT01631214/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT01631214/SAP_002.pdf